CLINICAL TRIAL: NCT02369198
Title: MesomiR 1: A Phase I Study of Intravenously Administered Epidermal Growth Factor Receptor -Targeted, EnGeneIC Delivery Vehicle (EDV)-Packaged, miR-16 Mimic (TargomiRs) for Patients With Malignant Pleural Mesothelioma (MPM) and Advanced Non-Small Cell Lung Cancer (NSCLC) Failing on Std Therapy
Brief Title: MesomiR 1: A Phase I Study of TargomiRs as 2nd or 3rd Line Treatment for Patients With Recurrent MPM and NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asbestos Diseases Research Foundation (Other)
Collaborators: EnGeneIC Limited (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HREC/13/CRGH/199
Record Dates: First submitted 2015-01-05; First posted 2015-02-23 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Malignant Pleural Mesothelioma; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Mesothelioma, Malignant; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm, open label TargomiRs (Experimental): TargomiRs are IV injected.
  Phase 1 Planned dose levels
  Dose level 1: 5 billion once a week Dose level 2: 5 billion twice a week Dose level 3: 5 billion once a week with cardiac monitoring Dose level 4: 2.5 billion twice a week with cardiac monitoring Dose level 5: as for dose level #3 with a dexamethasone challenge
  All patients begin on a micro dose of one billion and increase their dose over 2 weeks and reach their phase 1 dose level on week 3.
  Schedule of assessments includes laboratory and physical assessments in the 24 hours after each treatment as well as periodic assessments such as PET and CT scans for tumour assessment.
  100% of the data will be source data verified. Analysis will be simple phase 1 analysis based on a 3+3 model.
  Interventions: Drug: TargomiRs

INTERVENTIONS:
Drug: TargomiRs — TargomiRs are targeted minicells containing a microRNA mimic. They consist of three components: 1. A miR-16-based microRNA mimic. The miR-16 family has been implicated as a tumour suppressor in a range of cancer types. The mimic is a double-stranded, 23 base pair, synthetic RNA molecule. 2. Drug delivery vehicle - EDVs. EDVs are nonliving bacterial minicells (nanoparticles). They function as leak resistant micro-reservoir carriers that allow efficient packaging of a range of different drugs, proteins or nucleic acids. 3. Targeting moiety. The EDVs are targeted to EGFR-expressing cancer cells with an anti-EGFR bispecific antibody.
  TargomiRs are IV injected.

SUMMARY:
The first testing of TargomiRs in the human setting: dose-finding studies in patients with recurrent malignant pleural mesothelioma and non-small cell lung cancer

DETAILED DESCRIPTION:
TargomiRs are targeted minicells containing a microRNA mimic. They consist of three components: 1. A miR-16-based microRNA mimic. The miR-16 family has been implicated as a tumour suppressor in a range of cancer types. The mimic is a double-stranded, 23 base pair, synthetic RNA molecule. 2. Drug delivery vehicle - EDVs. EDVs are nonliving bacterial minicells (nanoparticles). They function as leak resistant micro-reservoir carriers that allow efficient packaging of a range of different drugs, proteins or nucleic acids. 3. Targeting moiety. The EDVs are targeted to EGFR-expressing cancer cells with an anti-EGFR bispecific antibody.

TargomiRs are IV injected.

Phase 1 Planned dose levels

Dose level 1: 5 billion once a week Dose level 2: 5 billion twice a week Dose level 3: 5 billion once a week with cardiac monitoring Dose level 4: 2.5 billion twice and week with cardiac monitoring Dose level 5: as above with an additional dexamethasone challenge

All patients begin on a micro dose of 1 billion once a week and escalate to the full phase 1 dose for their dose level on week 3.

Duration of treatment for each dose level is on a patient by patient basis. Officially the cycle is 8 weeks long however a patient can continue on treatment if they are deriving clinical benefit from the treatment.

If at any time point before or after the 8 week mark, a patient progresses, experiences ongoing or unreasonable toxicities or withdraws from the study, they will cease treatment.

Escalation of dose in cohorts of 3-6 patients per dose level. If at least 2 patients are observed to experience Dose Limiting Toxicity (DLT), the prior dose level is defined as the MTD.

Adherence to the protocol tends not to be problematic in patient groups where the trial treatment is their only treatment option. They are often very keen to participate and motivated to be part of the research.

ELIGIBILITY:
Inclusion Criteria:

Histological or cytological documentation of MPM or NSCLC and evidence of EGFR expression in tumour tissue.

Progression during or following the administration of standard 1st, 2nd or 3rd line therapy regimens.

Patient must have at least one measurable lesion according to the RECIST criteria version 1.1 for NSCLC and modified RECIST criteria for MPM

Male or female patients at least 18 years of age. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Life expectancy of at least 3 months.

Women of childbearing potential and men must agree to use adequate contraception from the time of signing of the informed consent form until at least 3 months after the last study drug administration.

Total bilirubin < 1.5 x the upper limit of normal (ULN) ALT and AST < 2.5 x ULN Amylase < 1.5 x ULN Serum creatinine < 1.5 x ULN GFR > 60 ml/min/m2 INR/PTT < 1.5 x ULN (patients who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists. Close monitoring with at least weekly evaluations will be performed until INR/APTT is stable (prior to administering the first dose)).

Platelet count > 100.000 and < 800.000, Hemoglobin (Hb) > 9 g/dl, Absolute Neutrophil count (ANC) > 1500/mm3. Alkaline phosphatase limit < 2.5 x ULN.

Exclusion Criteria:

Previous phase I drug treatment for the current diagnosis. Previous or concurrent cancer that is distinct in primary site or histology from MPM or NSCLC within 10 years from the date of screening EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumours (Ta, Tis and T1).

Presence of Salmonella antibodies. Herbal supplements (such as St John's Wort), nutritional supplements and also (multi)-vitamins taken within the last 30 days prior to dosing on Day 1 (and continued use, if appropriate), must be reviewed and approved by the local investigator.

Major surgical procedures in the last four weeks. Pregnancy or breast-feeding. Congestive heart failure > New York Heart Association (NYHA) class 2. Unstable angina (angina at rest) or new-onset angina (< 3 months). Myocardial infarction less than 6 months before eligibility screening.

Cardiac arrhythmias requiring anti-arrhythmic therapy (beta-blockers or digoxin are permitted).

Uncontrolled hypertension (Systolic blood pressure > 150 mmHg or diastolic pressure > 90 mm Hg despite optimal medical management).

Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including Transient Ischemic Attacks), deep vein thrombosis or pulmonary embolism within 6 months before the screening radiographic studies.

Ongoing infection > grade 2 NCI-CTCAE version 4.0 HIV infection. Chronic hepatitis B or C. Patients with a seizure disorder requiring medication. Symptomatic brain metastasis(es). The patient must not be undergoing acute steroid therapy or steroid tapering (Chronic steroid therapy is acceptable provided that the dose is stable for one month prior to and following screening radiographic studies).

Patients with a history of bleeding diathesis: Any hemorrhage or bleeding event of CTCAE Grade 3 within 4 weeks of the proposed start of study medication.

Renal failure requiring hemo-or peritoneal dialysis. Substance abuse, medical, psychological or social conditions that in the opinion of the investigator may interfere with the patient's participation in the study or evaluation of the study results.

Known hypersensitivity to bacterial proteins. Any medical condition that is unstable or could jeopardize the safety of the patient and his/her compliance in the study.

Unresolved toxicity higher than NCI-CTCAE (version 4.0) Grade 2 attributed to any prior therapy/procedure excluding alopecia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-09; Primary Completion 2017-01-04 (Actual); Study Completion 2017-01-04 (Actual)

PRIMARY OUTCOMES:
There is a composite primary outcome to establish maximum tolerated dose and dose limiting toxicities The MTD will be determined by the assessment of dose limiting toxicities. | DLTs assessed from treatment 1 for 2 weeks. MTD is measured from first treatment to toxicity (up to 18 months).
  There is a composite primary outcome to establish maximum tolerated dose and dose limiting toxicities.
  The MTD will be determined by the assessment of dose limiting toxicities. Toxicities, in the first 2 weeks of treatment for any given patient, are assessed with physical assessments 5 times in the 24 hours starting with a pre-dose assessment, and with laboratory assessments which are assessed 3 times in the 24 hours starting with pre-dose assessment.
  All adverse events are graded according to the CTCAE v4.0.
to evaluate the effect of multiple dosing of TargomiRs | the lab and physical assessments are conducted from first treatment, multiple times in a 24 hour period after treatment for up to 18 months
  to evaluate the effect of multiple dosing of TargomiRs using physical and lab assessments as well as tumour response via PET/CT.
to detect early signs of efficacy | 8 weeks, when formal assessment with RECIST is applied and QoL questionnaires assessed.
  to detect early signs of efficacy using QoL questionnaires and tumour response via PET/CT.

SECONDARY OUTCOMES:
QOL assessment | Baseline & weekly or twice weekly (depending on patient's cohort) up to 8 weeks
  QOL assessment using EORTC QLQ-C30 (Version 3)
ECOG PS change | ECOG PS will be assessed from baseline til 8 weeks
  to monitor changes in ECOG PS during treatment
Pulmonary function change | Pulmonary function is measured in screening and at 8 weeks
  to monitor pulmonary function parameters during treatment using FEV1 and Vital Capacity measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Nico vanZandwijk, PhD, Principal Investigator — University of Sydney
Locations (3):
- Australia (3):
  - Concord Repatriation General Hospital, Sydney, New South Wales
  - Chris O'Brien Lifehouse, Sydney, New South Wales
  - Northern Cancer Institute, Sydney, New South Wales

REFERENCES:
- [Result] Reid G, Pel ME, Kirschner MB, Cheng YY, Mugridge N, Weiss J, Williams M, Wright C, Edelman JJ, Vallely MP, McCaughan BC, Klebe S, Brahmbhatt H, MacDiarmid JA, van Zandwijk N. Restoring expression of miR-16: a novel approach to therapy for malignant pleural mesothelioma. Ann Oncol. 2013 Dec;24(12):3128-35. doi: 10.1093/annonc/mdt412. Epub 2013 Oct 22. PMID 24148817
- [Derived] Lucibello G, Mograbi B, Milano G, Hofman P, Brest P. PD-L1 regulation revisited: impact on immunotherapeutic strategies. Trends Mol Med. 2021 Sep;27(9):868-881. doi: 10.1016/j.molmed.2021.06.005. Epub 2021 Jun 26. PMID 34187739
- [Derived] van Zandwijk N, Pavlakis N, Kao SC, Linton A, Boyer MJ, Clarke S, Huynh Y, Chrzanowska A, Fulham MJ, Bailey DL, Cooper WA, Kritharides L, Ridley L, Pattison ST, MacDiarmid J, Brahmbhatt H, Reid G. Safety and activity of microRNA-loaded minicells in patients with recurrent malignant pleural mesothelioma: a first-in-man, phase 1, open-label, dose-escalation study. Lancet Oncol. 2017 Oct;18(10):1386-1396. doi: 10.1016/S1470-2045(17)30621-6. Epub 2017 Sep 1. PMID 28870611
- See also: Asbestos Diseases Research Institute — http://www.adri.org.au/